CLINICAL TRIAL: NCT07139041
Title: Treatment Strategy of Iparomlimab and Tuvonralimab Plus Chemotherapy for Inducing Conversion to Resectability in Initially Unresectable Stage III Non-Small Cell Lung Cancer: A Single-Arm Phase II Clinical Study
Brief Title: Iparomlimab and Tuvonralimab Plus Chemotherapy for Inducing Conversion to Resectability in Initially Unresectable Stage III NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Chen (Other)
Responsible Party: Sponsor-Investigator, Chang Chen, professor, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-NSCLC-QIBA-1004
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: NSCLC (Non-small-cell Lung Cancer)
Keywords: Iparomlimab and tuvonralimab;Conversion;Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and tuvonralimab plus chemotherapy (Other): Patients will receive Iparomlimab and tuvonralimab (5 mg/kg) plus chemotherapy (nab-paclitaxel, pemetrexed, or docetaxel) every 3 weeks.
  Interventions: Drug: Iparomlimab and tuvonralimab plus chemotherapy

INTERVENTIONS:
Drug: Iparomlimab and tuvonralimab plus chemotherapy — Squamous Cell Carcinoma: 2-4 cycles of Iparomlimab and tuvonralimab 5mg/kg Q3W (Day 1) + Albumin-bound Paclitaxel (100mg/m² Q3W D1/D8/D15 or130mg/m²D1/D8 or 260mg/m²D1) + Carboplatin (AUC=5) Q3W (D1) Non-Squamous Cell Carcinoma: 2-4 cycles of Iparomlimab and tuvonralimab 5mg/kg Q3W (D1) + Pemetrexed 500mg/m² Q3W (D1) + Carboplatin (AUC=5) Q3W (D1) Radical Chemoradiotherapy for Patients Unable to Undergo Surgery:Patients still unresectable after conversion therapy should start radical chemoradiotherapy within 6 weeks after the last conversion therapy dose. Chemoradiotherapy follows standard clinical practice, recommended as Cisplatin 30mg/m² QW (D1) + 60Gy radiotherapy.
  Adjuvant Therapy Phase:Iparomlimab and tuvonralimab 5mg/kg Q3W (D1) for up to 16 cycles.

SUMMARY:
This is a single-arm, multicenter Phase II clinical study designed to observe and evaluate the efficacy and safety of Iparomlimab and tuvonralimab plus chemotherapy in initially unresectable Stage III NSCLC. The study plans to enroll 69 Stage III NSCLC patients judged unresectable by a MDT team, with the R0 resection rate as the primary endpoint.

After completing 2-4 cycles of conversion therapy, the MDT team reassesses resectability. Subjects deemed suitable for surgical resection undergo surgery within 6 weeks after the last dose of conversion therapy. Subjects deemed unsuitable for surgery receive radical chemoradiotherapy, starting within 6 weeks after the last conversion therapy dose. Subjects unsuitable for both surgery and chemoradiotherapy will have their subsequent treatment decided by the project team.

Adjuvant therapy consists of Iparomlimab and tuvonralimab monotherapy (Q3W) for up to 16 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Signed an informed consent form
2. Patients aged ≥18
3. Histologically or cytologically confirmed Stage III (AJCC 9th ed.) squamous or non-squamous NSCLC (mixed tumors classified by predominant cell type), deemed unresectable by the MDT team based on at least one of the following criteria:

   1. Ipsilateral multi-station or confluent mediastinal lymph node metastasis: Imaging shows ipsilateral multi-station lymph node metastasis or confluent lymph node mass (>3cm diameter) or invasion of surrounding organs, making complete surgical clearance impossible.
   2. Contralateral or supraclavicular lymph node metastasis (N3): This includes contralateral hilar and mediastinal lymph node metastasis, or ipsilateral/contralateral supraclavicular lymph node metastasis.
   3. Invasion of vital organs or major vessels: Anatomical tumor or lymph node invasion directly involving the heart, major vessels (e.g., aorta, main pulmonary artery), trachea, esophagus, vertebral body (>50% involvement), or brachial plexus.
   4. Extensive chest wall and pleural invasion: Involvement of ribs, intercostal muscles, and chest wall soft tissues is extensive, requiring large chest wall resection that the patient's pulmonary function cannot tolerate, or impossible to clear surgically.
   5. Special anatomical location: e.g., superior sulcus tumor (Pancoast tumor) invading vertebrae/nerve plexus, recurrent laryngeal nerve involvement causing vocal cord paralysis, tumor extent precluding R0 resection.
   6. Patient unable to tolerate lobectomy or pneumonectomy: Insufficient cardiopulmonary reserve, severe cardiovascular disease, coagulation dysfunction, or other systemic diseases precluding lobectomy or pneumonectomy.
4. at least one measurable lesion according to RECIST 1.1 criteria
5. ECOG PS 0-1.
6. Pulmonary function must meet: FEV1 > 1.0 L and FEV1%> 40%
7. appropriate organ function

Exclusion Criteria:

1. NSCLC with small cell component identified on pathology (regardless of proportion); Histological types of large cell neuroendocrine carcinoma, sarcomatoid carcinoma, or NSCLC-NOS.
2. Known EGFR mutation or ALK rearrangement positivity (eligibility of subjects with other driver gene positivity will be determined by the project biomarker expert group).
3. Prior systemic anti-tumor therapy or thoracic radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
R0 Resection Rate | 2 years
  The proportion of patients who achieve complete tumor removal with no residual cancer cells at the surgical margin under microscopic examination after surgery

SECONDARY OUTCOMES:
2-year event-free survival (EFS) rate | 2 years
  The percentage of patients who remain free of disease progression, recurrence, or death within 24 months from the initiation of therapy
Pathologic Complete Response (pCR) | 2 years
  Pathologic complete response (pCR) rate is defined as the percentage of patients with no residual viable tumor cells in both primary tumor and sampled lymph nodes after neoadjuvant therapy